CLINICAL TRIAL: NCT04942262
Title: Identifying Diagnostic Criteria of Denture Adhesive Use in Complete Denture Wearers: A Quasi-experimental Study
Brief Title: Oral Health-related Quality of Life and Masticatory Function After Using Denture Adhesive and Denture Liner
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nareudee Limpuangthip, DDS, PhD, Dental staff at Department of Prosthodontics, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREC-DCU 2019-068
Record Dates: First submitted 2021-06-16; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Complete Denture; Complete Edentulism
Keywords: denture adhesive; oral impact; masticatory function; denture retention; denture stability
MeSH Terms: interventions — Dental Cements; Polident; halofantrine

STUDY DESIGN:
Intervention Model Description: Before and after intervention, and then allow the participants to decide whether to continue receiving the intervention
Masking Description: An external prosthodontist provided with a denture adhesive and knew who continued using denture adhesive.
  Meanwhile, the outcome assessor did not notice whether the participants continue using denture adhesive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- denture adhesive use (Experimental): Participants were instructed to use a cream-type denture adhesive (Polident®, GlaxoSmithKline, Ireland) once a day in the morning and use it throughout the day. They applied denture adhesive onto the tissue surface of their maxillary and mandibular dentures using a spot method. The participants had to remove the DA and clean the denture every day after the last meal by soaking and brushing the CD with liquid soap and a soft toothbrush under running tap water. Two gauze pads were used to remove DA from the denture and oral mucosa. After the 1-month trial period of DA use. The outcomes were evaluated with all participants using DA, and they had to choose whether they wanted to continue or discontinue using DA for another 1 month. At 1-month after continuing or discontinuing DA use. At this time, some participants used DA during the outcome evaluations, while some did not, depending on the patient's decision on DA use.
  Interventions: Drug: denture adhesive (Polident®, GlaxoSmithKline, Ireland)

INTERVENTIONS:
Drug: denture adhesive (Polident®, GlaxoSmithKline, Ireland) — cream-type denture adhesive available as an over-the-counter product in Thailand
  Other Names: Polident

SUMMARY:
80 complete denture (CD) wearers participated in the quasi-experimental study. Two outcomes were: 1) oral health-related quality of life (OHRQoL) assessed using the Oral Impacts on Daily Performances index, and 2) masticatory performance, determined by a peanut particle size after 20-stroke mastication. Denture retention and stability were evaluated using the Chulalongkorn University (CU)-modified Kapur method to classify the CD into acceptable or unacceptable quality. Data were collected at 3-time points: 1) at baseline (T0), 2) after a 1-month trial of denture adhesive (DA) use (T1), at which time the participants decided whether to continue using DA, and 3) 1-month after continued or discontinued using DA (T2).

DETAILED DESCRIPTION:
Participants The eligible participants were CD wearers randomly recruited from patients who visited the Prosthodontic clinic at the Faculty of Dentistry, Chulalongkorn University from 2015 to 2019. The inclusion criteria were patients who had worn removable maxillary and mandibular CDs for at least 6 months. The patients who wore a metal-based denture, had a history of DA use, had difficulty in responding to the interview, or were unwilling to follow the study protocol were excluded from the study.

Outcomes The primary outcome was OHRQoL determined using the Thai-version of Oral Impacts on Daily Performances index. The participants were interviewed whether they had difficulties in performing the following 8 daily activities: eat, speak, clean denture and mouth, sleep, smile, emotional stability, social contact, and carry out work or housework. The frequency and severity of each impact were rated using a five-point Likert scale, and their multiplication gave a condition-specific impact score. The overall oral impact score was the sum of all 8 activity scores. The prevalence of an oral impact was categorized into absence (score = 0) or presence of an oral impact (score > 0). The changes in oral impact score from T0 to T1 were categorized into 3 types: decreased (T0 score > T1 score), increased (T0 score < T1 score), and remained absent (T0 score = T1 score = 0).

The secondary outcome was masticatory performance assessed using the multiple sieve method of peanut mastication. The participants masticated 3 grams of roasted peanuts for 20 strokes in triplicate with a 15-minute resting interval between each test. The comminuted peanut particles were dried and sieved through 12 standard test sieves (Test sieve; Retcsh Technology GmbH) on a vibrating sieve shaker. A simple linear regression was plotted between the cumulative weight and diameter of each sieve test. The median peanut particle size (mm) was the sieve diameter through which 50% of the comminuted peanut particles passed. A smaller peanut particle size reflected a higher masticatory performance.

Intervention An external prosthodontist provided a cream-type DA (Polident®, GlaxoSmithKline, Ireland), and instructed the participants to use the DA cream once a day in the morning and use it throughout the day. They applied the DA onto maxillary and mandibular dentures on the tissue surface using a spot method. The participants had to remove the DA and clean the denture every day after the last meal by soaking and brushing the CD with liquid soap and a soft toothbrush under running tap water. Two gauze pads were used to remove DA from the denture and oral mucosa.

The OHRQoL, masticatory performance, and CD-quality were evaluated at 3-time points:

1. T0, at baseline before using the DA. The baseline information regarding the outcomes was evaluated. Then, the participants underwent a daily 1-month trial of DA use,
2. T1 (T0 + 1 month), after the 1-month trial period of DA use. The outcomes were evaluated with all participants using DA. The external prosthodontist asked the participants to choose whether they wanted to continue or discontinue using DA, and
3. T2 (T0 + 2 months), at 1-month after continuing or discontinuing DA use. At this time, some participants used DA during the outcome evaluations, while some did not, depending on the patient's decision on DA use.

A single-blind clinical trial protocol was created. One of the investigators (B.T.) performed the outcome assessment who did not notice whether the participants continue using DA.

ELIGIBILITY:
Inclusion Criteria:

* Wear removable maxillary and mandibular complete dentures for at least 6 months.

Exclusion Criteria:

* Wear a metal-based denture
* Have a history of DA use
* Unable to respond to the interview
* Unwilling to follow the study protocol.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life (OHRQoL) | 2 months
  The OHRQoL was assessed using the oral impacts on daily performances (OIDP) index. The participants were interviewed about whether they had difficulties in performing the following 8 daily activities within physical, psychological and social performances: eating, speaking and pronouncing, cleaning denture and mouth, sleeping, smiling, emotional stability, social contact, and carrying out work or housework. The frequency and severity of each impact were rated using a five-point Likert scale, and their multiplication gave a condition-specific (CS) impact score. The overall oral impact score was the sum of all 8 activity scores. The prevalence of an oral impact was categorized into absence (score = 0) or presence of an oral impact (score > 0).

SECONDARY OUTCOMES:
Masticatory performance using the multiple sieve method of peanut particle. | 2 months
  The participants masticated 3 grams of roasted peanuts for 20 strokes in triplicate with a 15-minute resting interval between each test. The comminuted peanut particles were dried and sieved through 12 standard test sieves (Test sieve; retch Technology GmbH) on a vibrating sieve shaker. A simple linear regression was plotted between the cumulative weight and diameter of each sieve test. The median peanut particle size (mm) was the sieve diameter through which 50% of the comminuted peanut particles passed. A smaller peanut particle size reflected a higher masticatory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nareudee Limpuangthip, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Dentistry, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limpuangthip N, Somkotra T, Arksornnukit M. Modified retention and stability criteria for complete denture wearers: A risk assessment tool for impaired masticatory ability and oral health-related quality of life. J Prosthet Dent. 2018 Jul;120(1):43-49. doi: 10.1016/j.prosdent.2017.09.010. Epub 2017 Nov 29. PMID 29195820
- [Result] Nicolas E, Veyrune JL, Lassauzay C. A six-month assessment of oral health-related quality of life of complete denture wearers using denture adhesive: a pilot study. J Prosthodont. 2010 Aug;19(6):443-8. doi: 10.1111/j.1532-849X.2010.00601.x. Epub 2010 Apr 29. PMID 20456031
- [Result] Ohwada G, Minakuchi S, Sato Y, Kondo H, Nomura T, Tsuboi A, Hong G, Itoh Y, Kawai Y, Kimoto S, Gunji A, Suzuki A, Suzuki T, Kimoto K, Hoshi N, Saita M, Yoneyama Y, Sato Y, Morokuma M, Okazaki J, Maeda T, Nakai K, Ichikawa T, Nagao K, Fujimoto K, Murata H, Kurogi T, Yoshida K, Nishimura M, Nishi Y, Murakami M, Hosoi T, Hamada T. Subjective Evaluation of Denture Adhesives: A Multicenter Randomized Controlled Trial. JDR Clin Trans Res. 2020 Jan;5(1):50-61. doi: 10.1177/2380084419837607. Epub 2019 Apr 11. PMID 30975019